CLINICAL TRIAL: NCT06391112
Title: Painting-Based Art of the Fetus During Non-Stress Testing Effect of Intervention on Maternal Anxiety and Fetal Parameters Randomized Controlled Clinical Trial
Brief Title: The Effect of Painting-Based Art Intervention on Maternal Anxiety and Fetal Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, CANSU AĞRALI, Research assistant, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OsmaniyeKAU-SBF-CA-01
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy Tests
Keywords: Art Therapy

STUDY DESIGN:
Intervention Model Description: There is a control and experimental group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Pregnant women in the control group will receive standard outpatient clinic treatment.
- Experimental group (Experimental): In the research, pregnant women in the Painting-Based Art Intervention group will be asked to imagine their own babies during the NST procedure and after imagining them, they will be asked to draw them in a drawing book.
  Interventions: Other: Painting Based Art intervention

INTERVENTIONS:
Other: Painting Based Art intervention — Painting Based Art Effect of Intervention on Maternal Anxiety and Fetal Parameters
  Arms: Experimental group

SUMMARY:
It is observed that art-based programs, one of the non-pharmacological methods, play an active role in improving the health and well-being of pregnant women and reducing anxiety, stress and depression. This shows that arts-based experiences offer women a unique opportunity to explore all dimensions of the transition to motherhood. When the literature is examined, it is seen that art-based interventions are used in birth units, neonatal intensive care and high-risk pregnancy units. However, no study has been found in which it was applied during the NST procedure. Therefore, the aim of our study is to examine the effect of picture-based art intervention on the fetus during the Non-Stress Test on maternal anxiety and fetal parameters.

DETAILED DESCRIPTION:
Hypotheses:

H1: Painting-Based Art Intervention positively affects NST results. H2: Painting-Based Art Intervention reduces the level of maternal anxiety.

Study protocol, methods and procedures to be applied:

Type of Research:

The research was planned as a randomized controlled clinical trial.

Place and Time of Research:

The research will be conducted at the NST polyclinic of Malatya Training and Research Hospital between January 2024 and May 2024.

Population and Sample of the Research The population of the research will consist of pregnant women who have applied to the NST polyclinic, have had at least one live birth, have had NST before, do not have any psychiatric or risky pregnancy diagnoses, do not have communication problems, and are older than the 32nd week of pregnancy.

There are 6 NST devices in the NST polyclinic where the research will be conducted. The assignment of pregnant women to the experimental and control groups will be made according to the device on which the NST procedure will be performed. It was decided by lottery method to perform the procedures on pregnant women in the experimental or control group with the devices numbered 1-6. In the draw held before the start of the research, it was determined that the pregnant women who would be included in the Painting-Based Art Intervention group with devices numbered 1, 4, 6, and the pregnant women who would be included in the control group with devices numbered 2, 3, 5 would undergo NST procedure. In order to prevent contamination between the experimental and control groups in the research, pregnant women who first form the control and then the experimental groups will be included in the study.

Criteria for inclusion in the study:

Not having any risk factors during pregnancy (preeclampsia, eclampsia, intrauterine growth retardation, PROM, gestational diabetes and hypertension, placenta previa, twin pregnancy, etc.).

Lack of uterine contraction, No cardiovascular disease diagnosed in the fetus, Pregnant women must be between the ages of 18-35 Conditions to be met before and during the NST procedure; Not having smoked or consumed alcohol at least two hours before the NST procedure, Having urinated before the NST procedure, Giving the pregnant woman the left side lateral position, Blood pressure values measured just before the NST procedure should be within the normal range,

Exclusion criteria for the study:

Any complications in the pregnancy, Any complications in the fetus, Refusal to accept the final test to be performed. Data Collection Process Data Collection Tools Data will be collected using the Introductory Information Form, State Anxiety Scale and Record Form for NST Findings, developed by the researchers using the literature.

Participant Introduction Form The Participant Introduction Form consists of questions that determine socio-demographic and obstetric characteristics, knowledge about NST findings, and drawing-based intervention.

NST Findings Record Form NST Findings Registration Form is a form used by researchers to evaluate NST results of pregnant women. This form contains data recording the findings of NST of pregnant women.

Evaluation of NST Findings Record Form; All pregnant women who agree to participate in the study will undergo NST with the NST device in the hospital. NST results of pregnant women will be evaluated by researchers.

As reactive NST; In the presence of at least two accelerations that last for at least 15 seconds and are 15 beats/minute more than the baseline beat within the 20-minute period during which the electronic fetal heart rate traces are printed, the result of the test will be considered as reactive NST.

As nonreactive NST; The absence of at least two accelerations that last for at least 15 seconds and are 15 beats/minute more than the baseline beat within the 20-minute period during which the electronic fetal heart rate traces are printed, in the presence of severe variable decelerations and late decelerations, or continuous fetal tachycardia of 160 beats/minute and above when the initial traces are normal. If it develops, the result will be evaluated as nonreactive NST.

State Anxiety Scale The state-trait anxiety scale, developed by Spielberg and his colleagues in 1964 to measure the anxiety levels of normal and abnormal individuals, was adapted into Turkish by Öner and Le Compte. The state anxiety part of the scale, which consists of two parts, will be used. There are 20 statements in both scales, and the answer options include four options, each ranging from 1 to 4.

The scales contain both direct (straight) expressions and reversed expressions. While direct expressions express negative emotions, tInverted expressions reflect positive emotions. In the State Anxiety Scale, these reversed statements are items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20. The statements in the scale are answered by selecting the options (1) not at all, (2) a little, (3) a lot and (4) completely in order to evaluate the emotions or behaviors according to the severity of the experiences. The total score obtained varies between 20 and 80, a high score indicates a high level of anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Not having any risk factors during pregnancy
* Lack of uterine contraction
* No cardiovascular disease diagnosed in the fetus
* Pregnant women must be between the ages of 18-35

Exclusion Criteria:

* Any complications in the pregnancy
* Any complications in the fetus
* Refusal to accept the final test to be performed

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
State Anxiety Scale | one week
  The state-trait anxiety scale, developed by Spielberg and his colleagues in 1964 to measure the anxiety levels of normal and abnormal individuals, was adapted into Turkish by Öner and Le Compte (1983). The state anxiety part of the scale, which consists of two parts, will be used. There are 20 statements in both scales and the answer options include four options, each ranging from 1 to 4.

SECONDARY OUTCOMES:
NST Findings Record Form | one week
  NST Findings Registration Form is a form used by researchers to evaluate NST results of pregnant women. This form contains data recording the NST findings of pregnant women.

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Nacar, Study Director — İnönü University
Locations (1):
- Turgut Özal Medical Training and Research Hospital, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No